CLINICAL TRIAL: NCT05807906
Title: The Effect of Virtual Reality Application on Fistula Puncture Associated Pain in Hemodialysis Patients
Brief Title: The Effect of Virtual Reality Application on Pain Due to Fistula Puncture in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Neşe Altinok Ersoy, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E1-22-2882
Record Dates: First submitted 2023-03-03; First posted 2023-04-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): virtual reality will be applied in the fistula puncture procedure in patients receiving hemodialysis treatment.
  Interventions: Other: virtual reality application
- Control Group (No Intervention): Routine nursing care and diet compliance narration

INTERVENTIONS:
Other: virtual reality application — The patient will continue to monitor the virtual reality application during the fistula puncture procedure.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to examine the effect of virtual reality application on fistula puncture-related pain (FPi-A) in hemodialysis patients.

Hypotheses of the Research:

H0-1: Virtual reality application has an effect on fistula puncture-related pain in HD patients.

H1-2: Virtual reality application has no effect on fistula puncture-related pain in HD patients.

In the study, virtual reality will be applied in the fistula puncture procedure in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
* Demographic/medical data will initially be recorded prior to fistula puncture.
* The patient will be prepared for the virtual reality application and fistula puncture and will be given a comfortable sitting position.
* Virtual reality glasses will be put on the patient 6 minutes before the fistula puncture and the application will be started.
* The patient will continue to monitor the virtual reality application during the fistula puncture procedure. It will be ensured that no communication with the patient is made until the application is finished.
* The application will be ended with the fixation of the needle on the fistula after the fistula puncture procedure.

ELIGIBILITY:
Inclusion Criteria:

* No diagnosis of neuropathic pain
* No sedatives, analgesics and sedatives are applied 3 hours before the application.
* Not taking recently taken antipsychotic drugs and tranquilizers,
* Deaf and visually impaired (to mark VAS pain)
* Without cognitive and psychiatric diagnosis
* Open to communication and cooperation
* Patients who agreed to participate in the study

Exclusion Criteria:

* Kidney transplant
* Discomfort due to virtual reality glasses
* Suspected/diagnosed COVID-19
* Patients who want to leave the study voluntarily
* Death
* Multiple fistula puncture attempts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Pain-VAS Scale | Assessing change of pain scores baseline, after each application for three weeks. Between third and fifth weeks any intervention will not be implemented and pain scale score will measure fifth week.
  VAS Scale is scored from 1 to 10. As the score increases, the severity of pain increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No